CLINICAL TRIAL: NCT03479437
Title: The TEMPO (Tracing the Effect of the MC4 Pathway in Obesity) Registry Involving Variants in Hypothalamic Genes Upstream or Downstream From the Melanocortin-4 Receptor (MC4R)
Brief Title: The TEMPO (Tracing the Effect of the MC4 Pathway in Obesity) Registry
Status: Completed | Type: Observational
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RM-493-020
Record Dates: First submitted 2018-03-12; First posted 2018-03-27 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Genetic Forms of Extreme Obesity
Keywords: Obesity; Melanocortin; TEMPO; MC4R; Genetic Obesity; hypothalamic; POMC; LEPR; PCSK1
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A voluntary prospective study that will allow registration and follow-up of individuals with MC4R pathway genetic obesity.

DETAILED DESCRIPTION:
Potential patients will be referred to coordinating centers by their healthcare provider (treating physician, diagnosing physician or primary care physician) and if eligible will be invited to enroll in the registry. The Registry Coordinating Center will be responsible for obtaining consent from adult patients and caregivers of minor patients (as well as assent from minors when appropriate), screening patients and enrolling them in the registry.

The registry will capture data entered by the patient, the patient's healthcare provider, and the patient's caregiver using online (electronic) survey tools administered at baseline, and annually thereafter. The patient's healthcare provider will complete the baseline Healthcare Provider survey tool, reporting the patient's baseline demographics, medical history, clinical information, and disease characteristics. The patient and caregiver will complete their dedicated baseline survey tools answering questions on the impact of disease on their everyday life. Survey tools include questions on patient and caregiver demographics, patient physical activity, patient food and hunger episodes, patient quality of life, and caregiver's perspective of disease burden on the family. Registry patients, caregivers, and healthcare providers will be contacted annually (approximately every 12 months) by the Registry Coordinating Center to complete an online follow-up survey tool including a smaller subset of questions from the baseline survey tools.

ELIGIBILITY:
Inclusion Criteria:

1. Extreme obesity patients aged 2 years and older.
2. Extreme obesity defined as:

   1. BMI > 40 kg/m2 in patients 18 years of age or older.
   2. BMI value that is >1.4 times the corresponding age/gender 95th percentile value in patients who are 2 through 17 years of age.
3. At least one of the following genotypes:

   1. Bi-allelic (homozygous or compound heterozygous) POMC, PCSK1, LEPR variants leading to the physician-confirmed diagnosis of either POMC or LEPR deficiency obesity.
   2. The presence of high-confidence, high-impact genetic variations (homozygote, compound heterozygote, heterozygote or composite heterozygote [i.e., heterozygous variants in more than a single gene]) in these same 3 genes (POMC, PCSK1 and LEPR) associated with the clinical presentation of extreme obesity
   3. The presence of other high-confidence, high-impact genetic variations (homozygote, compound heterozygote, heterozygote or composite heterozygote in the MC4R gene or other upstream MC4R-pathway genes and selected variants downstream in the MC4R-pathway (Table 1) that are carried by extreme obesity patients who do not demonstrate specific syndromic obesity clinical presentations. Selected Bardet-Biedl syndrome (BBS1 through BBS21) genetic variants or Alström syndrome (ALMS) genetic variants possibly contributing to non-syndromic forms of clinical extreme obesity will be eligible for enrollment.
4. Study participant and/or parent or caregiver can understand and comply with the requirements of the study, and able to understand and sign the written informed consent (IC)/assent, after being informed about the study.

Exclusion Criteria:

1. Patients with syndromic forms of obesity such as Bardet-Biedl syndrome or Alström syndrome. These patients will be referred to existing registries for these specific syndromic obesity (e.g., Clinical Registry in Bardet-Biedl syndrome [CRIBBS] for BBS patients).
2. Individual is, in the opinion of the study investigator, not suitable to participate in the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Extreme obesity in adults age 18 or older defined as a BMI >40 kg/m2 or subjects from age 2 through age 18 years with a BMI value that is >1.4 times the corresponding age/gender 95th percentile value will be eligible.
  Second, specific genotypic criteria involving defined major genes contributing to genetic obesity disorders will also be required for enrollment.
  Patients will be eligible to participate in the registry regardless of gender or geographic location. Other genetic forms of obesity may be added to this list as pathogenetic etiologies and the potential involvement of specific genes in the hypothalamus upstream or downstream of the MC4R become better understood.
  All known patients, or their caregivers, will be invited to participate. As new patients resulting from novel gene variants or defects are identified, registry patient enrollment will continue on an ongoing basis.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Quality of Life | 5 years
  Evaluate the quality of life through annual patient and caregiver reported surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Ihuoma Eneli, Principal Investigator — Nationwide Children's Hospital; Liz Stoner, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (2):
- Nationwide Children's Hospital, Columbus, Ohio, United States
- University of Alberta, Edmonton, Canada

IPD SHARING:
Plan to Share IPD: Undecided